CLINICAL TRIAL: NCT05234164
Title: HORIZON. Clinical Investigation of the Qmedics EXIST NiTi Stent Type FLEX & PULL in Adults With Peripheral Artery Disease (PAD)
Brief Title: HORIZON Prospective Clinical Investigation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Qmedics AG (Industry)
Collaborators: Policlinico di Monza (Unknown); University Clinical Hospital of Bialystok (Unknown); University Hospital, Catania (Other); Erasmus Medical Center (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120884
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Disease
Keywords: stenotic lesions; Peripheral Arterial Disease; occluded lesions; Superficial Femoral Artery; nitinol stent; self-expanding stent; Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Subjects requiring treatment of the SFA will undergo a calcification review based on the Fanelli classification. Subjects graded with Fanelli 1 or 2, and subjects requiring treatment of the P1 segment of the proximal popliteal artery will be treated with the Exist 6F NiTi Stent type FLEX.
  Subject graded with Fanelli 3 and 4 will be treated with the Exist 6F NiTi Stent PULL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXIST 6F NiTi Stent System FLEX (Experimental): Stent implantation of lesions in the SFA graded with Fanelli 1 and 2, and lesions in the P1 segment of the proximal popliteal artery.
  Interventions: Device: EXIST 6F NiTi Stent System FLEX
- EXIST 6F NiTi Stent System PULL (Experimental): Stent implantation of lesions in the SFA graded with 3 and 4.
  Interventions: Device: EXIST 6F NiTi Stent System PULL

INTERVENTIONS:
Device: EXIST 6F NiTi Stent System FLEX — Subjects requiring treatment of the P1 segment of the proximal popliteal artery will be treated with the Exist 6F NiTi Stent FLEX type. Subjects requiring treatment of the SFA will undergo an additional calcification review based on the Fanelli classification. Subjects graded with Fanelli 1 or 2 will be treated with the Exist 6F NiTi Stent FLEX type.
  Arms: EXIST 6F NiTi Stent System FLEX
Device: EXIST 6F NiTi Stent System PULL — Subjects requiring treatment of the SFA will undergo a calcification review based on the Fanelli classification. Subjects graded with Fanelli grade 3 and 4 will be treated with the Exist 6F NiTi Stent PULL type.
  Arms: EXIST 6F NiTi Stent System PULL

SUMMARY:
The objective of this clinical investigation is to demonstrate and provide long term clinical data on safety and performance of the Exist 6F NiTi stent system type FLEX & PULL in a prospective investigation for the treatment of adult patients with de novo or re-stenotic symptomatic atherosclerotic lesions in Peripheral Artery Disease (PAD) requiring treatment of the Superficial Femoral Artery (SFA) or Proximal Popliteal Artery (P1 segment).

DETAILED DESCRIPTION:
This is a multicenter, prospective study with clinical and radiographic follow-up for 24 months months post-procedure. Approximately two hundred thirty subjects will be enrolled (115 subjects will receive the FLEX type and 115 subjects the PULL type) in several centers, minimum 10 patients per investigational center. All patients will be evaluated at 30 days and 6-, 12- and 24-months post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

- Clinical:

1. Patient age 18 years or older
2. Subject is willing and able to provide consent before any study specific test or procedure is performed, signs the consent form, and agrees to attend all required follow-up visits
3. Symptoms of peripheral arterial disease classified as Rutherford Category 2, 3 or 4 or Fontaine Class IIb or III
4. The stenotic or occlusive lesion in Superficial Femoral Artery (SFA) and proximal popliteal artery, P1 segment, is considered suitable for stenting
5. No underlying medical condition is present which would prevent the subject from performing the required testing or from completing the study.
6. Stable medical condition

   * Anatomical criteria:
7. Included TASC II, A-B-C measured on pre- angio CT-scan (if CT-scan is standard of care)
8. Lesions must be one or multiple that can be treated with maximum two stents, maximum one overlapping and maximum length of the stent 25 cm
9. Patent ipsilateral iliac, popliteal (P2 and P3) and at least one tibial vessel

Exclusion Criteria:

- Clinical criteria:

1. Subjects pregnant, breastfeeding or planning to become pregnant during the trial participation
2. Documented life expectancy less than 24 months due to other medical co-morbid condition(s)
3. Thrombophlebitis or deep vein thrombosis within the past 30 days.
4. Unable to assume DAPT (Dual Antiplatelet Therapy)
5. Concomitant renal failure with serum creatinine level > 2.5 mg/dL (or > 220 µmol/L) or GFR < 30 ml/min/1,73 m2
6. Unresolved neutropenia (white blood cell count < 3,000 / µL) or thrombocytopenia (platelet count < 80,000 / µL) at the time of the index procedure
7. Unresolved bleeding disorder (INR ≥ 1.2) at the time of the index procedure
8. Active gastrointestinal bleeding
9. Anticoagulation therapy for other medical condition

   * Anatomical criteria:
10. Target lesion(s) received previous treatment within 30 days prior to enrolment (point of enrolment is defined as the time when the trial device enters the body)
11. Previously stented ipsilateral SFA
12. Prior peripheral vascular bypass surgery involving the target limb(s)
13. Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion
14. Target lesion requires the use of cutting balloons, atherectomy or drug coated balloons (DCB) during the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Primary patency | 12 months
  The primary patency rate (defined as freedom from more than ≥ 50% restenosis) at 12 months post-procedure as measured by Peak Systolic Velocity ratio (PSVr) assessed with Duplex ultrasound (DUS). A PSVr ≥ 2,5 suggests a reduction in the luminal diameter >50%.
Major Adverse Events | 1 month
  Freedom from procedure- or stent-related Major Adverse Events (MAEs) at 30-days post index-procedure will be reported. MAE is defined as all causes of death and target limb major amputation, defined as amputation of the lower limb at the ankle level or above.

SECONDARY OUTCOMES:
Improvement of Rutherford / Fontaine classification | 6- and 12-months
  Clinical success Defined as improvement of Rutherford / Fontaine classification of one class or more as compared to the pre-procedure and an ankle-brachial index improvement (ABI) by ≥ 0.15.
Primary patency | 12-months
  Compare the Exist 6F NiTi stent primary patency with >50% of subjects with peripheral artery disease with literature data.
Rate of stent fracture | 12- and 24-months
  Stent fracture rate is evaluated with x-ray. Stent fracture is defined according to classification on x-ray.
Freedom from Target Lesion Revascularization | 1 month, 6-, 12- and 24-months
  Defined as the absence of revascularization (by any means) of the target lesion (fTLR).
Walking and mobility | 1 month, 6-, 12- and 24-months
  Improvement of walking and mobility is assessed by change in the 36-Item Short Form Survey (SF-36) score from baseline.
Patency rate | 24 months
  Patency rate as measured by Peak Systolic Velocity ratio (PSVr) assessed with Duplex ultrasound (DUS). A PSVr ≥ 2,5 suggests a reduction in the luminal diameter >50%.
Major Adverse Events | 24 months
  Procedure- or stent-related Major Adverse Events (MAEs) post index-procedure will be reported. MAE is defined as all causes of death and target limb major amputation, defined as amputation of the lower limb at the ankle level or above.

OTHER OUTCOMES:
Self-reported Quality of life | 1 month, 6-, 12- and 24-months
  Improvement of quality of life is assessed by change in the 36-Item Short Form Survey (SF-36) score from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Patteet, MD, Study Director — Qmedics AG
Locations (2):
- University Hospital of Catania, Catania, Sicily, Italy
- University Clinical Hospital of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No